CLINICAL TRIAL: NCT06800378
Title: The Impact of the Sedative-Hypnotic Medication Zolpidem on Performance in Road Cycling
Brief Title: Zolpidem's Effects on Road Cycling Performance
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan Normal University (Other)
Collaborators: Ten-Chen General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 113-A-01-02
Record Dates: First submitted 2024-12-23; First posted 2025-01-30 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Healthy
MeSH Terms: interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Other): 10 mg starch
  Interventions: Other: Placebo
- Drug (Experimental): 10 mg Zolpidem
  Interventions: Drug: Zolpidem 10 mg

INTERVENTIONS:
Drug: Zolpidem 10 mg — Zolpidem tartrate 10 mg tablet (taken before bedtime)
  Arms: Drug
Other: Placebo — Starch 10 mg tablet (taken before bedtime)
  Arms: Placebo

SUMMARY:
This study will recruit 15 healthy participants who regularly engage in cycling as their primary physical activity. Recruitment will take place at the hospital, where participants will sign an informed consent form and complete a health survey. The experiments will be conducted at the Exercise Physiology Laboratory in Gongguan, National Taiwan Normal University. Participants will need to familiarize themselves with the procedures before the formal tests. Prior to the measurements, participants must complete: (1) a Sleep Quality Questionnaire and (2) a Sleep Pattern Questionnaire.

This study follows a double-blind design and involves two formal experiments. Two weeks before the experiments, participants will complete forms regarding sleep quality, recent Functional Threshold Power (FTP) over the past 1-2 months, and will receive an explanation of the study. One week before the experiments, participants will visit Dr. Kuo-Yi Weng at the Rheumatology and Immunology Clinic of Zhongli Ten-Chan Hospital to obtain the study medication, Zolpidem .

On the evening before the first experiment, participants will report to the laboratory before 7:00 PM. At 8:59 PM, they will be randomly assigned to take either 10 mg of Zolpidem or a placebo. At 9:00 PM, participants will go to bed wearing a sleep monitoring device (Fitbit Charge 4). At 4:00 AM, they will wake up, complete the Leeds Sleep Evaluation Questionnaire (Self-reported), and have breakfast. The formal experiment will begin at 5:00 AM, during which participants will use the Zwift online platform to simulate a 60-kilometer ride to measure athletic performance. The two formal experiments will be spaced one week apart.

DETAILED DESCRIPTION:
1. Specimen Collection:

1. On the test day, arm tissue glucose levels will be collected using continuous glucose monitoring (CGM), which will continue until the experiment concludes.
2. Fingerstick blood samples will be taken using a lancet to measure glucose and lactate levels at 0,10,20,40,50 and 60 kilometers.

2. Prohibitions, Restrictions, and Requirements for Participants During the Trial:

1. Training and Sleep Patterns: Participants are required to maintain their usual training routines and sleep patterns without changing their schedules increasing training intensity. This is to control for changes in physical performance and sleep quality during the trial period.
2. Diet: Participants should consume the same or similar foods the day before and the day of the trial to minimize the impact of dietary changes on the experiment. 3.Restrictions: Participants are prohibited from consuming caffeinated beverages such as tea, coffee, or energy drinks on the night before and the morning of the trial to avoid potential interference with the results.

ELIGIBILITY:
Inclusion Criteria:

* Adults over 20 years old
* Bicycle age over 2 years
* Rides more than twice a week
* Does not regularly use sedative-hypnotic drugs or first-generation antihistamines that aid in sleep
* Does not have drinking or smoking habits (≤1 time per week)
* Has competition experience (has participated in cycling competitions over 100 kilometers or other cycling races)
* Has used an indoor bicycle trainer
* Average sleep time is between 11:00 PM and 1:00 AM

Exclusion Criteria:

* Irregular sleep and shift workers
* Individuals with medical, psychiatric, and sleep disorders

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2024-06-26 (Actual); Primary Completion 2024-12-22 (Actual); Study Completion 2024-12-29 (Actual)

PRIMARY OUTCOMES:
Physiological Indicator (Lactate) for 40km at 70%FTP | Approximately 1 to 1.5 hours during each study intervention.
  Lactate in mmol/L .Testing will be conducted using an indoor trainer (TACX NEO) to assess whether taking medication affects lactate changes.Lactate will be collected at 10, 20, 30, 40 kilometers, respectively. A total of four times.
Physiological Indicator (Blood Glucose) for 40km at 70%FTP | Approximately 1 to 1.5 hours during each study intervention.
  Glucose in mg/dL . Testing will be conducted using an indoor trainer (TACX NEO) to evaluate whether taking medication affects blood glucose changes.The evaluation will be conducted when the participants complete 10, 20, 30, and 40 km of cycling(Using CGM). A total of four times.
Rate of Perceived Exertion for 40 km at 70% FTP | Approximately 1 to 1.5 hours during each study intervention.
  Borg Scale (6-20) .Testing will be conducted using an indoor trainer (TACX NEO) to determine whether taking medication influences changes in the Rate of Perceived Exertion (RPE).The evaluation will be conducted when the participants complete 10, 20, 30, and 40 km of cycling. A total of four times.
20KM Time Trial | Approximately 30 to 60 min during each study intervention.
  Time trial (minute) .Testing will be conducted using an indoor trainer (TACX NEO) to assess whether taking medication affects the time trial (TT) performance.Participants performed a 20 km time trial (TT) after completing 40 km at 70% FTP, and the completion time was recorded.A total of one times.
Average Power for 20KM Time Trial | Approximately 30 to 60 min during each study intervention.
  Average Power(W).Testing will be conducted using an indoor trainer (TACX NEO) to evaluate whether taking medication affects the average power output.Participants performed a 20 km time trial (TT) after completing 40 km at 70% FTP, and the average power was recorded.A total of one times.
Physiological Indicator (Blood Glucose) for 20KM Time Trial | Approximately 30 to 60 min during each study intervention.
  Glucose in mg/dl . Testing will be conducted using an indoor trainer (TACX NEO) to assess whether taking medication affects blood glucose changes during the time trial.The evaluation will be conducted when the participants complete 10, 20 km of Time Trial. A total of two times.
Physiological Indicator (Lactate) for 20KM Time Trial | Approximately 30 to 60 minutes during each study intervention.
  Testing will be conducted using an indoor trainer (TACX NEO) to evaluate whether taking medication affects lactate changes during the time trial.The evaluation will be conducted when the participants complete 10, 20 km of Time trial . A total of two times .
Rate of Perceived Exertion for 20km Time trial | Approximately 30 to 60 minutes during each study intervention.
  RPE：Borg Scale (Score：6-20 ).Testing will be conducted using an indoor trainer (TACX NEO) to determine whether taking medication influences changes in the Rate of Perceived Exertion (RPE) during the time trial.The evaluation will be conducted when the participants complete 10, 20 km of Time trial . A total of two times .
Sleep Duration (Minutes) | The monitoring duration is 7 hours during each study intervention.
  Sleep Duration in Minutes.Sleep duration will be measured using Fitbit Charge 4 to evaluate the differences in sleep length between taking and not taking medication.Measurements will begin after taking medication at 9:00 PM and conclude upon waking up the next day at 4:00 AM. Sleep duration will be recorded using Fitbit Charge 4.
Sleep Latency (Minutes): | The monitoring duration is 7 hours during each study intervention.
  Sleep latency in minutes . Sleep latency will be measured using Fitbit Charge 4 to evaluate the differences in the time taken to fall asleep between taking and not taking medication.Measurements will begin after taking medication at 9:00 PM and conclude upon waking up the next day at 4:00 AM. Sleep potency will be recorded using Fitbit Charge 4.

CONTACTS AND LOCATIONS:
Locations (1):
- Ten-Chan General hospital, Taoyuan District, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wilms B, Chamorro R, Hallschmid M, Trost D, Forck N, Schultes B, Molle M, Sayk F, Lehnert H, Schmid SM. Timing Modulates the Effect of Sleep Loss on Glucose Homeostasis. J Clin Endocrinol Metab. 2019 Jul 1;104(7):2801-2808. doi: 10.1210/jc.2018-02636. PMID 30807636
- [Background] Temesi J, Arnal PJ, Davranche K, Bonnefoy R, Levy P, Verges S, Millet GY. Does central fatigue explain reduced cycling after complete sleep deprivation? Med Sci Sports Exerc. 2013 Dec;45(12):2243-53. doi: 10.1249/MSS.0b013e31829ce379. PMID 23760468
- [Background] Saner NJ, Lee MJ, Kuang J, Pitchford NW, Roach GD, Garnham A, Genders AJ, Stokes T, Schroder EA, Huo Z, Esser KA, Phillips SM, Bishop DJ, Bartlett JD. Exercise mitigates sleep-loss-induced changes in glucose tolerance, mitochondrial function, sarcoplasmic protein synthesis, and diurnal rhythms. Mol Metab. 2021 Jan;43:101110. doi: 10.1016/j.molmet.2020.101110. Epub 2020 Oct 31. PMID 33137489
- [Background] Rosenberg RP, Hull SG, Lankford DA, Mayleben DW, Seiden DJ, Furey SA, Jayawardena S, Roth T. A randomized, double-blind, single-dose, placebo-controlled, multicenter, polysomnographic study of gabapentin in transient insomnia induced by sleep phase advance. J Clin Sleep Med. 2014 Oct 15;10(10):1093-100. doi: 10.5664/jcsm.4108. PMID 25317090
- [Background] Papanikolaou DD, Astara K, Vavougios GD, Daniil Z, Gourgoulianis KI, Stavrou VT. Elements of Sleep Breathing and Sleep-Deprivation Physiology in the Context of Athletic Performance. J Pers Med. 2022 Mar 2;12(3):383. doi: 10.3390/jpm12030383. PMID 35330382
- [Background] Mougin F, Simon-Rigaud ML, Davenne D, Renaud A, Garnier A, Kantelip JP, Magnin P. Effects of sleep disturbances on subsequent physical performance. Eur J Appl Physiol Occup Physiol. 1991;63(2):77-82. doi: 10.1007/BF00235173. PMID 1748108
- [Background] Leong RLF, Cheng GH, Chee MWL, Lo JC. The effects of sleep on prospective memory: A systematic review and meta-analysis. Sleep Med Rev. 2019 Oct;47:18-27. doi: 10.1016/j.smrv.2019.05.006. Epub 2019 May 31. PMID 31216498
- [Background] Horoszok L, Baleeiro T, D'Aniello F, Gropper S, Santos B, Guglietta A, Roth T. A single-dose, randomized, double-blind, double dummy, placebo and positive-controlled, five-way cross-over study to assess the pharmacodynamic effects of lorediplon in a phase advance model of insomnia in healthy Caucasian adult male subjects. Hum Psychopharmacol. 2014 May;29(3):266-73. doi: 10.1002/hup.2395. PMID 24911577
- [Background] Holgado D, Manresa-Rocamora A, Zamboni L, Lugoboni F, Peiro AM, Zandonai T. The effect of benzodiazepines on exercise in healthy adult participants: A systematic review. J Addict Dis. 2022 Jul-Sep;40(3):336-344. doi: 10.1080/10550887.2021.1990640. Epub 2021 Nov 9. PMID 34751107
- [Background] Haraldsdottir K, Sanfilippo J, McKay L, Watson AM. Decreased Sleep and Subjective Well-Being as Independent Predictors of Injury in Female Collegiate Volleyball Players. Orthop J Sports Med. 2021 Sep 9;9(9):23259671211029285. doi: 10.1177/23259671211029285. eCollection 2021 Sep. PMID 34527756
- [Background] Grobler LA, Schwellnus MP, Trichard C, Calder S, Noakes TD, Derman WE. Comparative effects of zopiclone and loprazolam on psychomotor and physical performance in active individuals. Clin J Sport Med. 2000 Apr;10(2):123-8. doi: 10.1097/00042752-200004000-00007. PMID 10798794
- [Background] Gramaglia E, Ramella Gigliardi V, Olivetti I, Tomelini M, Belcastro S, Calvi E, Dotta A, Ghigo E, Benso A, Broglio F. Impact of short-term treatment with benzodiazepines and imidazopyridines on glucose metabolism in healthy subjects. J Endocrinol Invest. 2014 Feb;37(2):203-6. doi: 10.1007/s40618-013-0016-y. Epub 2014 Jan 9. PMID 24497220
- [Background] Craven J, McCartney D, Desbrow B, Sabapathy S, Bellinger P, Roberts L, Irwin C. Effects of Acute Sleep Loss on Physical Performance: A Systematic and Meta-Analytical Review. Sports Med. 2022 Nov;52(11):2669-2690. doi: 10.1007/s40279-022-01706-y. Epub 2022 Jun 16. PMID 35708888
- [Background] Collomp K, Fortier M, Cooper S, Long A, Ahmaidi S, Prefaut C, Wright F, Picot M, Cote MG. Performance and metabolic effects of benzodiazepine during submaximal exercise. J Appl Physiol (1985). 1994 Aug;77(2):828-33. doi: 10.1152/jappl.1994.77.2.828. PMID 8002535
- [Background] Chase JD, Roberson PA, Saunders MJ, Hargens TA, Womack CJ, Luden ND. One night of sleep restriction following heavy exercise impairs 3-km cycling time-trial performance in the morning. Appl Physiol Nutr Metab. 2017 Sep;42(9):909-915. doi: 10.1139/apnm-2016-0698. Epub 2017 May 3. PMID 28467857
- [Background] Boonstra TW, Stins JF, Daffertshofer A, Beek PJ. Effects of sleep deprivation on neural functioning: an integrative review. Cell Mol Life Sci. 2007 Apr;64(7-8):934-46. doi: 10.1007/s00018-007-6457-8. PMID 17347797
- [Background] Azboy O, Kaygisiz Z. Effects of sleep deprivation on cardiorespiratory functions of the runners and volleyball players during rest and exercise. Acta Physiol Hung. 2009 Mar;96(1):29-36. doi: 10.1556/APhysiol.96.2009.1.3. PMID 19264040